CLINICAL TRIAL: NCT04735224
Title: Long-term Risks After Endoscopic Retrograde Cholangiopancreatography (ERCP) With Sphincterotomy.
Brief Title: Complications After Endoscopic Retrograde Cholangiopancreatography
Acronym: ERCP
Status: Completed | Type: Observational
Sponsor: Juan Carlos Martín del Olmo (Other)
Responsible Party: Sponsor-Investigator, Juan Carlos Martín del Olmo, MD, PhD. Associate Profesor Valladolid University, Hospital Medina del Campo
Organization: Hospital Medina del Campo (Other)
Other Study IDs: HMCampo2
Record Dates: First submitted 2020-12-22; First posted 2021-02-03 (Actual); Last update posted 2021-02-03 (Actual); Status verified 2021-01

CONDITIONS: Choledocholithiasis With Acute Cholangitis (Diagnosis); Acute Pancreatitis Due to Gallstones
Keywords: ERCP; ERCP complications; Endoscopic Sphincterotomy
MeSH Terms: conditions — Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Retrospective study to analyze benign complications and malignancy risks after ERCP with sphincterotomy. All patients who received a ERCP with sphincterotomy for a benign disease will be included. Post-ERCP hepato-biliary complications in the follow-up will be registered.

DETAILED DESCRIPTION:
This is a single center retrospective study. All patients that received an ERCP with sphincterotomy for a benign disease from 1995 will be included.

The exclusion criteria are diagnosis of primary malignant tumors in the liver, bile ducts including peri-ampullary region and pancreas in the ERCP. Loss of follow-up less than two years after the ERCP and biliopancreatic malignancy diagnostic in this period. The initial work-up included laboratory test, ultrasound scan and, when precise, computed tomography (CT) and magnetic resonance image (MRI).

The data collected will be:

1. Age, sex, comorbidities, long of hospital stay.
2. ERCP indications.
3. ERCP sphincterotomy or precut, biliary stent insertion and type of stent.
4. post-ERCP diagnosis, abnormal diameter of biliary tree.
5. ERCP repetition and causes.
6. Immediate complications like bleeding, residual choledocholithiasis, ascending cholangitis, pancreatitis, and cholecystitis, and their number after more than two months.
7. Malignant complications after more than two years: cholangiocarcinoma, hepatocarcinoma and ductal pancreatic adenocarcinoma.

Stistical analyses will be performed using SPSS, ver. 25.0 (SPSS Inc., Chicago Illinois, USA). The demographics, perioperative data, operation details, length of hospital stay, morbidity, mortality and pathologic and oncological outcomes are expressed as numbers and percentages for qualitative variables and medians and interquartile ranges (IQRs) for quantitative variables.

Univariate and multivariate logistic regression analyses will be employed to determine the risk factors for the development short-term and long-term complications. Variables with P<0.1 in the univariate analysis will be further introduced into the multivariate analysis with the Wald selection method. P values < 0.05 were considered statistically significant.

This study involved the use of data from clinical records. To guarantee the proper handling of the information, the data were treated confidentially and anonymously according to the provisions of the Spanish Organic Law 15/1999, of 13 December 1999, on Personal Data Protection (LOPD). All methods were performed in accordance with the guidelines and regulations established by the Declaration of Helsinki (1964, revised in 1983) on biomedical research in humans, the Spanish Royal Decree 1090/2015, of December 4, which regulates clinical trials with drugs, the Research Ethics Committees with drugs and the Spanish Registry of Clinical Studies. Ethical approval from the Clinical Trials and Ethics Committee of Valladolid University was granted.

ELIGIBILITY:
Inclusion Criteria:

* Patients having undergone ERCP with sphincterotomy for benign diseases between 1995 and 2015

Exclusion Criteria:

* Diagnosis of primary malignant tumors in the liver, bile ducts including ampullary region, and pancreas in the ERCP test.
* Patients with follow-up less than two years after the ERCP and biliopancreatic malignancy diagnostic in this period.

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Patients having undergone ERCP with sphincterotomy for benign diseases between 1995 and 2015
Sampling Method: Non-Probability Sample
Enrollment: 500 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2020-10-10 (Actual); Study Completion 2020-12-20 (Actual)

PRIMARY OUTCOMES:
long-term complications after ERCP with sphincterotomy | 10 years
  Long- terms complications registered

SECONDARY OUTCOMES:
characteristics of patients who develop complications after endoscopy sphincterotomy | 10 years
  defined characteristics

OTHER OUTCOMES:
association between ERCP with sphincterotomy and the development of neoplasm in the bile ducts | 10 years
  risks of malignancy

CONTACTS AND LOCATIONS:
Overall Officials: Juan Carlos Martin Del Olmo, MD, PhD, Study Director — Hospital Medina del Campo; Mercedes Ibáñez García, MD, PhD, Principal Investigator — Hospital Medina del Campo; Carlos Guijarro, MD, PhD, Study Chair — Hospital Medina del Campo; Kostantin Shirai, MD, PhD, Study Chair — Hospital Medina del Campo; Cristina López Mestanza, MD, PhD, Study Chair — Hospital Medina del Campo

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] McCune WS, Shorb PE, Moscovitz H. Endoscopic cannulation of the ampulla of vater: a preliminary report. Ann Surg. 1968 May;167(5):752-6. doi: 10.1097/00000658-196805000-00013. No abstract available. PMID 5646296
- [Background] Nakajima M, Kimoto K, Fukumoto K, Ikehara H, Kawai K. Endoscopic sphincterotomy of the ampulla of Vater and removal of common duct stones. Am J Gastroenterol. 1975 Jul;64(1):34-43. No abstract available. PMID 1155423
- [Background] Oliveira-Cunha M, Dennison AR, Garcea G. Late Complications After Endoscopic Sphincterotomy. Surg Laparosc Endosc Percutan Tech. 2016 Feb;26(1):1-5. doi: 10.1097/SLE.0000000000000226. PMID 26679684
- [Background] ASGE Standards of Practice Committee; Chathadi KV, Chandrasekhara V, Acosta RD, Decker GA, Early DS, Eloubeidi MA, Evans JA, Faulx AL, Fanelli RD, Fisher DA, Foley K, Fonkalsrud L, Hwang JH, Jue TL, Khashab MA, Lightdale JR, Muthusamy VR, Pasha SF, Saltzman JR, Sharaf R, Shaukat A, Shergill AK, Wang A, Cash BD, DeWitt JM. The role of ERCP in benign diseases of the biliary tract. Gastrointest Endosc. 2015 Apr;81(4):795-803. doi: 10.1016/j.gie.2014.11.019. Epub 2015 Feb 7. No abstract available. PMID 25665931
- [Background] ASGE Standards of Practice Committee; Chandrasekhara V, Khashab MA, Muthusamy VR, Acosta RD, Agrawal D, Bruining DH, Eloubeidi MA, Fanelli RD, Faulx AL, Gurudu SR, Kothari S, Lightdale JR, Qumseya BJ, Shaukat A, Wang A, Wani SB, Yang J, DeWitt JM. Adverse events associated with ERCP. Gastrointest Endosc. 2017 Jan;85(1):32-47. doi: 10.1016/j.gie.2016.06.051. Epub 2016 Aug 18. No abstract available. PMID 27546389
- [Background] Sung JY, Leung JW, Shaffer EA, Lam K, Olson ME, Costerton JW. Ascending infection of the biliary tract after surgical sphincterotomy and biliary stenting. J Gastroenterol Hepatol. 1992 May-Jun;7(3):240-5. doi: 10.1111/j.1440-1746.1992.tb00971.x. PMID 1611012

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-03-22): https://cdn.clinicaltrials.gov/large-docs/24/NCT04735224/Prot_SAP_000.pdf